CLINICAL TRIAL: NCT00002395
Title: An Open, Comparative Phase II Study of Immediate Versus Delayed Treatment With Topotecan HCl Given as a Continuous 21-Day Infusion Every 28 Days to Patients With AIDS-Related Progressive Multifocal Leukoencephalopathy
Brief Title: Safety and Effectiveness of Topotecan HCl to Treat HIV-Infected Patients With AIDS-Related Progressive Multifocal Leukoencephalopathy (PML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SmithKline Beecham (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 284A; Protocol 111; SK&F 104864-A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: HIV Infections; Leukoencephalopathy, Progressive Multifocal
Keywords: AIDS-Related Opportunistic Infections; Leukoencephalopathy, Progressive Multifocal; Infusions, Intravenous; Drug Administration Schedule; Topotecan
MeSH Terms: conditions — HIV Infections; Leukoencephalopathy, Progressive Multifocal; AIDS-Related Opportunistic Infections | interventions — Topotecan

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
The purpose of this study is to see if it is safe and effective to give topotecan through a vein to treat HIV-infected patients with PML, an opportunistic (AIDS-related) infection caused by a virus that infects brain tissue and causes damage to the brain and the spinal cord.

Topotecan fights HIV and the JC virus (the virus that causes PML) in laboratory experiments.

DETAILED DESCRIPTION:
Topotecan, a cytotoxic DNA topoisomerase-I inhibitor that crosses the blood-brain barrier, inhibits the replication of JC virus (the virus that causes PML) in vitro, at concentrations that are not toxic to human cells. Topotecan also inhibits the replication of HIV-1 and the function of Tat (which upregulates the replication of JC virus).

Patients are randomized to be treated immediately with topotecan or to have treatment delayed for 8 weeks. The dosing schedule for patients receiving immediate or delayed treatment is topotecan as a continuous 21-day intravenous infusion every 28 days. All patients must have received optimal, stable antiretroviral therapy for 3 weeks prior to entry and preferably will continue that therapy during the study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have PML, including symptoms of PML.
* Are able to complete the study.
* Agree to have a catheter inserted in a vein.
* Have taken at least 3 weeks of a stable anti-HIV drug combination (unless they are unable to take anti-HIV drugs).
* Are at least 18 years old.
* Agree to use effective methods of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history of certain central nervous system (CNS) diseases.
* Have a history of certain psychiatric disorders, such as bipolar disorder or schizophrenia.
* Have syphilis that has not been treated.
* Have certain severe medical problems, including AIDS-related opportunistic infections (such as PCP) that require treatment.
* Have received chemotherapy in the past 30 days.
* Have ever received chemotherapy for PML.
* Are pregnant or breast-feeding.
* Are taking certain medications, including any other investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Veteran's Administration Hosp / West LA, Los Angeles, California
  - HIV Institute / Davies Med Ctr, San Francisco, California
  - Univ of Miami, Miami, Florida
  - Johns Hopkins Univ, Baltimore, Maryland
  - Albany Med College / Div of HIV Medicine, Albany, New York